CLINICAL TRIAL: NCT02231268
Title: Observational Study Via Internet to Assess a 6-months Treatment With GLADEM
Brief Title: Observational Study to Assess a 6-months Treatment With Gladem
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 533.2
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Sertraline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Depressive patients
  Interventions: Drug: Gladem

INTERVENTIONS:
Drug: Gladem

SUMMARY:
* Evaluation of a 6-months treatment with Gladem
* Experiences with the internet for performing a postmarketing study (PMS) trial

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years old
* De novo prescription of Gladem
* Treatment with Gladem intended for at least 6 months
* Depressive disorders

Exclusion Criteria:

* Known hypersensitivity against sertraline
* Concomitant treatment with monoamine oxidase (MAO)-inhibitors, selegiline, moclobemide (washout for at least 14 days necessary)
* Concomitant treatment with other serotoninergic substances like tryptophan or fenfluramine
* Instable epilepsy

According to product information (October 1998) Gladem prescription was possible with precautions in the following cases:

* Patients with stable epilepsy
* Patients with restricted liver functions
* Suicidal patients
* Patients in emotional state and marked sleeping disorders

According to product information (October 1998) Gladem should only be prescribed during pregnancy and lactation period, if the expected benefit was greater than the risk. Women of childbearing age should use Gladem only in combination with sufficient contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: out-patients
Enrollment: 546 (Actual)
Dates: Start 2000-09; Primary Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Scale (HAMD-6) | 3 months, 6 months

SECONDARY OUTCOMES:
Global assessment of efficacy on a 4-point scale | up to 6 months
Global assessment of compliance on a 4-point scale | up to 6 months
Global assessment of tolerability on a 4-point scale | up to 6 months
Clinical global impression score | up to 6 months
Number of responders | up to 6 months
  >= 50 % reduction in HAMD-6 score
Change in HAMD subscores | baseline, 6 months
Number of patients with adverse drug reactions | up to 6 months